CLINICAL TRIAL: NCT05642312
Title: A Phase III, Multicenter, Randomized, Double-Masked, Sham-Controlled Study to Investigate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Vamikibart Administered Intravitreally in Patients With Uveitic Macular Edema
Brief Title: A Study to Investigate Vamikibart in Participants With Uveitic Macular Edema
Acronym: Meerkat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GR44277; 2022-501793-19-00 (EU CTIS Number)
Record Dates: First submitted 2022-12-06; First posted 2022-12-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Uveitic Macular Edema
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Participants will receive 4 high-dose vamikibart intravitreal (IVT) injections every 4 weeks (Q4W) to Week 12, followed by as-needed (PRN) dosing from Week 20 to Week 48.
  Interventions: Drug: Vamikibart
- Arm B (Experimental): Participants will receive 4 low-dose vamikibart IVT injections Q4W to Week 12, followed by PRN dosing from Week 20 to Week 48.
  Interventions: Drug: Vamikibart
- Arm C (Sham Comparator): Participants will receive 4 sham injections Q4W to Week 12, followed by PRN sham dosing from Week 20 to Week 48.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Vamikibart — Participants will receive vamikibart IVT injection
  Other Names: RO7200220
  Arms: Arm A; Arm B
Other: Sham — Participants will receive a sham procedure that mimics an IVT injection.
  Arms: Arm C

SUMMARY:
This study will assess the efficacy and safety of vamikibart in participants with uveitic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Female participants: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception as defined by the protocol
* Diagnosis of macular edema associated with non-infectious uveitis (NIU)
* Diagnosis of active or inactive, acute, or chronic NIU of any etiology and of any anatomical type (anterior, intermediate, posterior, panuveitis)
* BCVA letter score of 73 to 19 letters (inclusive) on Early Treatment Diabetic Retinopathy Study (EDTRS)-like charts

Exclusion Criteria:

* Evidence of active or latent syphilis infection
* Evidence of active or latent tuberculosis infection and/or positive tuberculosis assay, or previous or current HIV diagnosis
* Serious acute or chronic medical or psychiatric illness
* History of major ocular and non-ocular surgical procedures
* Uncontrolled IOP or glaucoma or chronic hypotony
* Any anatomical changes or media opacity in the study eye preventing evaluation of retina, vitreous, and capture of study images
* Prior use of IVT biologics including anti-VEGFs less than 2-4 months prior to Day 1; received IVT Methotrexate within 4 months prior to Day 1
* Prior macular laser therapy, cataract surgery within 6 months and laser capsulotomy within 3 months of Day 1
* Topical corticosteroids and/or topical NSAID > 3 drops per day in the 14 days prior to Day 1 (D1); intraocular or periocular corticosteroid injections in the 2 months prior to D1; subconjunctival corticosteroid injection within 1 month prior to Day 1; an OZURDEX implant in the 4 months prior to D1; YUTIQ, RETISERT or ILUVIEN implant in the 3 years prior to D1
* Diagnosis of macular edema due to any cause other than NIU
* Any major ocular conditions that may require medical or surgical intervention during the study period to prevent vision loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with ≥ 15 letter improvement from baseline in best-corrected visual acuity (BCVA) at Week 16 | Week 16

SECONDARY OUTCOMES:
Proportion of participants with ≥ 15 letter improvement from baseline in BCVA at Week 20 | Week 20
Change from baseline in BCVA at Week 16 | Week 16
Change from baseline in central subfield thickness (CST) at Week 16 | Week 16
Change from Baseline in BCVA at Weeks 20 and 52 | Weeks 20 and 52
Change from baseline in CST at Weeks 20 and 52 | Weeks 20 and 52
Proportion of participants with uveitic macular edema secondary to non-infectious uveitis (UME) resolution defined by standardized (by machine) CST threshold <325um on optical coherence tomography (OCT) from baseline at Weeks 16 and 52 | Weeks 16 and 52
Time to rescue treatment | Up to Week 52
Number of rescue treatments received | Up to Week 52
Type of rescue treatments received | Up to Week 52
Proportion of participants with ≥15 letter improvement from baseline in BCVA at Week 16 and 52 | Weeks 16 and 52
Proportion of participants without ≥15 letter loss from baseline in BCVA at Week 16 and 52 | Weeks 16 and 52
Number of PRN injections received | Up to Week 52
Time to first PRN injection | Up to Week 52
Change from baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) at Weeks 16 and 52 | Weeks 16 and 52
Percentage of participants with ocular adverse events (AEs) | Up to Week 52
Percentage of participants with non-ocular AEs | Up to Week 52
Percent change from baseline in corneal endothelial cell density at Week 24 | Week 24
Percentage of participants with adverse events of special interest (AESIs) | Up to Week 52
Percent change from baseline in corneal endothelial cell density at Week 52 | Week 52
Aqueous humor (AH) concentration of vamikibart | Up to Week 52
Serum concentration of vamikibart | Up to Week 52
Anti-drug antibody titer to vamikibart | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (77):
- United States (16):
  - Kaiser Permanente Southern California, Los Angeles, California
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - VitreoRetinal Surgery, PLLC., Minneapolis, Minnesota
  - Truhlsen Eye Institute, Omaha, Nebraska
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Wake Forest Baptist Health Eye Centre, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Investigational Drug Services, Columbus, Ohio
  - Oregon Health & Science Uni, Portland, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Tennessee Retina PC, Nashville, Tennessee
  - Austin Clinical Research LLC, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
- Austria (3):
  - LKH-Univ.Klinikum Graz, Graz
  - Kepler Universitätskliniken GmbH - Med Campus III, Linz
  - Medizinische Universitat Wien, Vienna
- Brazil (4):
  - Retina Clinic, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESPX, São Paulo, São Paulo
  - CEMAPE - Centro Médico, São Paulo, São Paulo
  - Fiocruz - Fundação Oswaldo Cruz, Rio de Janeiro
- Canada (3):
  - Kensington Vision and Research Centre, Toronto, Ontario
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec
- China (10):
  - Peking Union Medical College Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - Shanghai First People's Hospital, Shanghai
  - Tianjin Medical University Eye Hospital, Tianjin
  - Eye Hospital, Wenzhou Medical University, Wenzhou
  - Ren Min Hospital Affiliated Wu Han University, Wuhan
- Israel (7):
  - Rambam Medical Center, Haifa
  - Hadassah MC, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin MC, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky MC, Tel Aviv
  - Assuta Hashalom Medical Center, Tel Aviv
- Italy (4):
  - AUSL ? IRCCS Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - ASL 4 SSR Ospedale Santa Maria di Montallegro, Rapallo, Liguria
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Asst Fatebenefratelli Sacco, Milan, Lombardy
- Hospital de la Ceguera APEC, Mexico City, Mexico CITY (federal District), Mexico
- Netherlands (2):
  - Het Oogziekenhuis Rotterdam, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (5):
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddzia? Kliniczny Okulistyki i Onkologii Okulistycznej, Krakow
  - SPSK nr 1 w Lublinie, Lublin
  - SPEKTRUM Osrodek Okulistyki Klinicznej, Wroclaw
- Portugal (3):
  - AIBILI - Association for Innovation and Biomedical Research on Light, Coimbra
  - Instituto de Oftalmologia Dr. Gama Pinto, Lisbon
  - Hospital de Santa Maria, Lisbon
- South Korea (9):
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Ajou University Medical Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Kim's Eye Hospital, Seoul
- Taiwan (3):
  - Taipei Veterans General Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- United Kingdom (7):
  - Queen Elizabeth Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Bristol Eye Hospital, Bristol
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucestershire
  - Royal Liverpool University Hospital, Liverpool
  - Western Eye Hospital, London
  - James Cook Hospital, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing